CLINICAL TRIAL: NCT06220890
Title: Clinical Performance of Two Different Bevel Preparations in Class IV Lesions Using Nanofilled Composite: A Randomized Clinical Study
Brief Title: Clinical Performance of Two Different Bevel Preparations in Class IV Lesions Using Nanofilled Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Akankshya Behera
Record Dates: First submitted 2024-01-13; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Class IV Dental Caries
MeSH Terms: interventions — Tooth Preparation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Class IV lesion with 2 mm bevel (BV) (Experimental): All the enamel margins will be beveled at a 45-degree angle of the width of approximately 2 mm, enamel selectively etched, bonding of tooth using universal adhesive will be done and restored with nano-filled composite.
  Interventions: Procedure: Tooth preparation in Class IV lesions with 2mm bevel
- Class IV lesion with 2mm stair-step chamfer (SSC) (Experimental): Enamel margins facially will be prepared 2mm deep in stair-step chamfer form, enamel selectively etched, and bonding of tooth using universal adhesive will be done and restored with nano-filled composite.
  Interventions: Procedure: Tooth preparation in Class IV lesions with 2mm stair-step chamfer

INTERVENTIONS:
Procedure: Tooth preparation in Class IV lesions with 2mm bevel — Class IV cavity with 2 mm bevel will be restored with nano-filled composite and clinical performance will be evaluated based on FDI criteria.
  Arms: Class IV lesion with 2 mm bevel (BV)
Procedure: Tooth preparation in Class IV lesions with 2mm stair-step chamfer — Class IV cavity with 2 mm stair step chamfer will be restored with nano-filled composite and clinical performance will be evaluated based on FDI criteria.
  Arms: Class IV lesion with 2mm stair-step chamfer (SSC)

SUMMARY:
The purpose of the study is to compare and evaluate clinical performance between two different bevel preparations in Class IV lesions using nano-filled composite restorations.

DETAILED DESCRIPTION:
The main reason for failure in anterior composite restorations is restoration fracture and aesthetic appearance. Restorations in anterior teeth are subjected to high-impact stresses produced through an incisal angle in class IV restorations, require high fracture resistance. It is the biomechanics of restorations that determine their functionality, retention, and functional longevity. Stair-step chamfer preparation is a modification of chamfer preparation that follows the vertical and horizontal anatomical contours, hence, achieves high degree of aesthetics along with exposure of enamel for bonding. According to current literature, no studies have analyzed the clinical performance of different bevel design using direct nano-filled composite resin restorations in Class IV lesions.

Therefore, the aim of this study is to compare and evaluate clinical performance between two different bevel preparations in Class IV lesions using nano-filled composite restorations.

Study will be conducted at Post Graduate Institute of Dental Sciences, Rohtak in Department of Conservative Dentistry & Endodontics. Time Frame of the study will be 12 months. Patients ≥ 18 years of age with Class IV lesion in maxillary central incisor, lateral incisor due to fracture or primary/ recurrent caries will be enrolled in the study.

After complete carious removal, tooth will be prepared in class IV lesions according to 2mm bevel or 2mm stair-step chamfer preparation group, selective enamel etching and bonding of the tooth using universal adhesive will be done. The cavity will be restored using nanofilled composite by layering technique. The restorations will be undergoing the standard finishing and polishing procedures.

Follow up of patients will be carried out at 3 months for clinical evaluation, 6 and 12 months for both radiographic and clinical evaluation. Restorations will be assessed clinically according to FDI criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age at the time of treatment.
* Class IV lesion in maxillary central incisor, lateral incisor due to fracture or primary/ recurrent caries.
* Patients with complete and normal occlusion and teeth with proximal contacts.
* Patients not having periodontal or pulpal diseases.
* Positive response to the cold test and electric pulp test.

Exclusion Criteria:

* Patients with immunocompromised status or debilitating systemic diseases.
* Patients with uncontrolled parafunctional habits.
* Class IV lesion with involvement of pulp.ix
* Class IV lesions with no involvement of dentin.
* Patients presenting extremely poor oral hygiene.
* Patient with high caries index

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of 2 mm bevel and stair step chamfer in Class IV lesions using nanofilled composite restorations. | 12 months
  Evaluation of Clinical and radiographic success of class IV lesions with 2mm bevel and stair step chamfer with nanofilled composite restorations will be assessed by FDI criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sanjay Tewari, MDS, Study Director — POSTGRADUATE INSTITUTE OF DENTAL SCIENCE,ROHTAK ,HARYANA,INDIA,124001
Locations (1):
- PGIDS, Rohtak, Haryana, India